CLINICAL TRIAL: NCT02548156
Title: Intra-oral Kinetics of Fluoride Containing Dentifrices in a Modified Saliva Clearance Study
Brief Title: Intra Oral Kinetics of Fluoride Containing Dentifrices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 204777
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Tooth Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test dentifrice (Other): 1.5g (± 0.05g) of Test dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse
  Interventions: Other: Test Dentifrice; Other: Orange Juice; Other: De-ionised water
- Reference dentifrice (Other): 1.5g (± 0.05g) of Reference dentifrice followed by 10mL of de-ionised water rinse, then 10 mL water rinse
  Interventions: Other: Reference Dentifrice; Other: De-ionised water
- Comparator dentifrice (Other): 1.5g (± 0.05g) of Comparator dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse
  Interventions: Other: Comparator Dentifrice; Other: Orange Juice; Other: De-ionised water

INTERVENTIONS:
Other: Test Dentifrice — Marketed dentifrice containing 1150ppm fluoride and 5% w/w KNO3
  Arms: Test dentifrice
Other: Reference Dentifrice — Marketed dentifrice containing 1150ppm fluoride and 5% w/w KNO3
  Arms: Reference dentifrice
Other: Comparator Dentifrice — Marketed dentifrice containing 1150ppm fluoride and 5% w/w KNO3
  Arms: Comparator dentifrice
Other: Orange Juice — Teeth will be rinsed with orange juice followed by rinsing with de-ionised water in test dentifrice and comparator dentifrice arms.
  Arms: Comparator dentifrice; Test dentifrice
Other: De-ionised water — Teeth will be rinsed with de-ionised water followed by reference dentifrice and followed by rinsing with orange juice in test dentifrice and comparator dentifrice arms.

SUMMARY:
The aim of this study is to assess the impact of formulation differences on fluoride retention clearance with US levels of fluoride (1150 ppm of fluoride) by evaluating and comparing between treatments the concentrations of fluoride and calcium ions in saliva over 60 minutes after a single brushing with US marketed fluoridated dentifrices and following a dietary acid challenge post 60 minutes of brushing with study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Aged 18-65 years
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general and mental health with, in the opinion of the investigator or medically qualified designee:

  1. No clinically significant and relevant abnormalities of medical history or oral examination
  2. Absence of any condition that would impact on the participant's safety or well being or affect the individual's ability to understand and follow study procedures and requirements
* A minimum of 20 permanent natural teeth
* A gum-base stimulated whole saliva flow rate ≥ 0.8 mL/min and an unstimulated whole saliva flow rate ≥ 0.5 mL/min.

Exclusion Criteria:

* Pregnant or breast feeding women
* Presence of chronic debilitating disease.
* Any condition that causes xerostomia as determined by the Investigator.
* Evidence of untreated caries.
* Gross periodontal disease.
* Tongue or lip piercing or presence of dental implants. Professional tooth cleaning or dental treatment during study. Oral surgery or extraction within 6 weeks of the screening visit.
* Self reported oral symptoms including lesions, sores or inflammation
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Currently taking antibiotics or have taken antibiotics within 2 weeks of the screening visit
* Any medication that could affect salivary flow or cause xerostomia as determined by the Investigator
* Use of multivitamins, calcium supplements and or fluoride supplements within 7 days of treatment phase
* Participant unwilling to abstain from smoking for at least 4 hours on the day of each test visit
* Recent history (within the last year) of alcohol or other substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ellesmere Port, Cheshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one Centre United Kingdom.
Pre-assignment Details: A total of 59 participants were screened, out of which 29 were randomized. Of the 29 randomized participants, 28 completed the study.
Groups:
- Sequence 1: Test/Comparator/Reference: Dentifrice: Firstly 1.5g (± 0.05g) of Test dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; secondly 1.5g (± 0.05g) of Comparator dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; thirdly 1.5g (± 0.05g) of Reference dentifrice followed by 10mL of de-ionised water rinse, then 10 mL DI water rinse were given to participants in Period 1, Period 2 and Period 3 respectively. Each period was separated by washout period of 7+/-1 day.
- Sequence 2: Test/Reference/Comparator: Dentifrice: Firstly 1.5g (± 0.05g) of Test dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; secondly 1.5g (± 0.05g) of Reference dentifrice followed by 10mL of de-ionised water rinse, then 10 mL DI water rinse; thirdly 1.5g (± 0.05g) of Comparator dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse were given to participants in Period 1, Period 2 and Period 3 respectively. Each period was separated by washout period of 7+/-1 day.
- Sequence 3: Comparator/Test/Reference: Dentifrice: Firstly 1.5g (± 0.05g) of Comparator dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; secondly 1.5g (± 0.05g) of Test dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; thirdly 1.5g (± 0.05g) of Reference dentifrice followed by 10mL of de-ionised water rinse, then 10 mL DI water rinse were given to participants in Period 1, Period 2 and Period 3 respectively. Each period was separated by washout period of 7+/-1 day.
- Sequence 4: Comparator/Reference/Test: Dentifrice: Firstly 1.5g (± 0.05g) of Comparator dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; secondly 1.5g (± 0.05g) of Reference dentifrice followed by 10mL of de-ionised water rinse, then 10 mL DI water rinse; thirdly 1.5g (± 0.05g) of Test dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse were given to participants in Period 1, Period 2 and Period 3 respectively. Each period was separated by washout period of 7+/-1 day.
- Sequence 5: Reference/Test/Comparator: Dentifrice: Firstly 1.5g (± 0.05g) of Reference dentifrice followed by 10mL of de-ionised water rinse, then 10 mL DI water rinse; secondly 1.5g (± 0.05g) of Test dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; thirdly 1.5g (± 0.05g) of Comparator dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse were given to participants in Period 1, Period 2 and Period 3 respectively. Each period was separated by washout period of 7+/-1 day.
- Sequence 6: Reference/Comparator/Test: Dentifrice: Firstly 1.5g (± 0.05g) of Reference dentifrice followed by 10mL of de-ionised water rinse, then 10 mL DI water rinse; secondly 1.5g (± 0.05g) of Comparator dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse; thirdly 1.5g (± 0.05g) of Test dentifrice followed by 10mL of de-ionised water rinse, then 10 mL orange juice rinse were given to participants in Period 1, Period 2 and Period 3 respectively. Each period was separated by washout period of 7+/-1 day.
Period: Period 1
Arm/Group | Sequence 1: Test/Comparator/Reference: Dentifrice | Sequence 2: Test/Reference/Comparator: Dentifrice | Sequence 3: Comparator/Test/Reference: Dentifrice | Sequence 4: Comparator/Reference/Test: Dentifrice | Sequence 5: Reference/Test/Comparator: Dentifrice | Sequence 6: Reference/Comparator/Test: Dentifrice
Started | 5 | 5 | 4 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1: Test/Comparator/Reference: Dentifrice | Sequence 2: Test/Reference/Comparator: Dentifrice | Sequence 3: Comparator/Test/Reference: Dentifrice | Sequence 4: Comparator/Reference/Test: Dentifrice | Sequence 5: Reference/Test/Comparator: Dentifrice | Sequence 6: Reference/Comparator/Test: Dentifrice
Started | 5 | 5 | 4 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence 1: Test/Comparator/Reference: Dentifrice | Sequence 2: Test/Reference/Comparator: Dentifrice | Sequence 3: Comparator/Test/Reference: Dentifrice | Sequence 4: Comparator/Reference/Test: Dentifrice | Sequence 5: Reference/Test/Comparator: Dentifrice | Sequence 6: Reference/Comparator/Test: Dentifrice
Started | 5 | 5 | 4 | 5 | 4 | 5
Completed | 5 | 5 | 4 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1: Test/Comparator/Reference: Dentifrice | Sequence 2: Test/Reference/Comparator: Dentifrice | Sequence 3: Comparator/Test/Reference: Dentifrice | Sequence 4: Comparator/Reference/Test: Dentifrice | Sequence 5: Reference/Test/Comparator: Dentifrice | Sequence 6: Reference/Comparator/Test: Dentifrice
Started | 5 | 5 | 4 | 5 | 4 | 5
Completed | 5 | 5 | 4 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: Test/Comparator/Reference: Dentifrice | Sequence 2: Test/Reference/Comparator: Dentifrice | Sequence 3: Comparator/Test/Reference: Dentifrice | Sequence 4: Comparator/Reference/Test: Dentifrice | Sequence 5: Reference/Test/Comparator: Dentifrice | Sequence 6: Reference/Comparator/Test: Dentifrice
Started | 5 | 5 | 4 | 5 | 4 | 5
Completed | 5 | 5 | 4 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All the participants randomized in this study.
Arm/Group | Overall Study
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (9.12)
Gender [Count of Participants; unit: Participants]
  Female | 23
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Fluoride Ions in Saliva 60 Minutes Post Brushing Prior to Administration of the Orange Juice or De-ionised Water Rinse
Description: Concentration of fluoride ions in saliva at 60 minutes after a single brushing with a fluoride dentifrice prior to rinsing with either de-ionised (DI) water or orange juice (OJ). Descriptive data is presented as least square (LS) mean and standard error (SE). SE for Fluoride is the SE of the raw mean.
Time Frame: 60 minutes
Population: The Per Protocol (PP) population was a subset of the ITT population (All randomized participants who had received study treatment and have at least one post-baseline efficacy measurement). n= number of participants analyzed for this outcome.
Measure: Least Squares Mean (Standard Error); unit: parts per million(ppm)
Arm/Group | Test Dentifrice | Reference Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 28 | 28 | 28
parts per million(ppm) | 0.23 (0.0469) | 0.23 (0.0430) | 0.15 (0.0485)
Statistical Analysis 1: Comparison: Test Dentifrice vs Reference Dentifrice vs Comparator Dentifrice; Test and Reference dentifrice combined vs. Comparator dentifrice; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANCOVA of log transformed data: subject (random), treatment (fixed) and period (fixed) as factors, participant-level baseline and period-level baseline minus participant-level baseline as covariates; Ratio of LS mean = 1.52 — Treatment difference from ANCOVA of log transformed data. This therefore represents the ratio of the first named treatment to the second named treatment. A ratio >1 favors the first named treatment

2. Secondary Outcome: Concentrations of Fluoride and Calcium Ions in Saliva Post Brushing Prior to Administration of Orange Juice or De-ionised Water Rinse
Description: Concentration of fluoride and calcium ions in saliva at baseline, 1, 5, 10, 15, 30 and 60 minutes (for calcium only) after a single brushing with a fluoride dentifrice
Time Frame: up to 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Test Dentifrice | Reference Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 28 | 28 | 28
ppm
  Fluoride: At baseline (n=26, 28, 26) | 0.045 (0.0125) | 0.032 (0.0084) | 0.031 (0.0072)
  Fluoride: At 1 minute (n=27, 28, 26) | 8.775 (0.8301) | 8.794 (1.0562) | 7.630 (0.7497)
  Fluoride: At 5 minute (n=27, 27, 27) | 3.881 (0.4115) | 4.132 (0.4759) | 3.492 (0.4664)
  Fluoride: At 10 minute (n=26, 26, 26) | 1.831 (0.1980) | 1.951 (0.2654) | 1.476 (0.1524)
  Fluoride: At 15 minute (n=27, 27, 26) | 1.346 (0.1827) | 1.188 (0.1550) | 0.942 (0.1432)
  Fluoride: At 30 minute (n=26, 27, 27) | 0.656 (0.1065) | 0.600 (0.0810) | 0.479 (0.0723)
  Calcium: At Baseline (n=26, 25, 22) | 29.749 (0.9428) | 28.357 (1.0162) | 28.661 (1.0657)
  Calcium: At 1 minute (n=23, 28, 25) | 28.300 (1.5171) | 27.217 (1.0689) | 14.931 (1.0999)
  Calcium: At 5 minute (n=16, 17, 22) | 27.818 (1.3743) | 26.070 (1.4638) | 17.227 (0.9170)
  Calcium: At 10 minute (n=16, 16, 21) | 27.472 (1.0061) | 25.672 (1.1944) | 20.133 (1.0395)
  Calcium: At 15 minute (n=18, 20, 20) | 28.319 (1.0783) | 27.227 (0.8656) | 23.761 (1.2803)
  Calcium: At 30 minute (n=17, 18, 20) | 28.650 (1.0725) | 27.323 (1.0325) | 24.196 (1.3196)
  Calcium: At 60 minute (n=23, 20, 22) | 28.198 (1.0073) | 27.094 (1.0560) | 27.104 (1.3777)

3. Secondary Outcome: Concentrations of Fluoride and Calcium Ions in Saliva Following Administration of the Orange Juice or De-ionised Water Rinse
Description: Concentration of fluoride and calcium ions in saliva following a rinse with either de ionised water or OJ 60 minutes after a single brushing with a fluoride dentifrice
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ppm
Arm/Group | Test Dentifrice | Reference Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 28 | 28 | 28
ppm
  Fluoride Ion concentration(n=27, 28, 27) | 0.349 (0.0349) | 0.169 (0.1104) | 0.277 (0.1601)
  Calcium Ion concentration (n=26, 22, 25) | 15.015 (4.3355) | 27.263 (4.7113) | 14.805 (4.0473)

4. Secondary Outcome: Concentrations of Fluoride and Calcium Ions in the Initial Expectorate, De-ionised Water Rinse Post Brushing Expectorate, and 60 Minutes Post Brushing Following Administration of Orange Juice or De-ionised Water Rinse
Description: Concentration of fluoride and calcium ions in the initial expectorate, de-ionized water rinse post brushing expectorate, and 60 minutes post brushing following administration of orange juice or de-ionised water rinse
Time Frame: up to 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Test Dentifrice | Reference Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 28 | 28 | 28
ppm
  Fluoride: In initial expectorate | 178.522 (61.1593) | 168.728 (54.3780) | 164.708 (54.2632)
  Fluoride: Post-Brushing De-Ionised Water Rinse Ex | 8.377 (4.2346) | 7.721 (4.1721) | 7.443 (3.4546)
  Fluoride: 60 Minutes Post Brushing | 0.166 (0.0609) | 0.046 (0.0370) | 0.135 (0.0563)
  Calcium: In initial expectorate | 17.096 (4.7864) | 17.467 (4.1241) | 2.500 (0.0000)
  Calcium: Post-Brushing De-Ionised Water Rinse Ex | 4.959 (2.2712) | 4.438 (2.2141) | 2.500 (0.0000)
  Calcium: 60 Minutes Post Brushing | 96.165 (9.2357) | 4.600 (2.0507) | 99.189 (17.2771)

ADVERSE EVENTS:
Arm/Group | Test Dentifrice | Reference Dentifrice | Comparator Dentifrice
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 8/28 | 3/29 | 5/28
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (N=28) | Reference Dentifrice (N=29) | Comparator Dentifrice (N=28)
Chapped Lips (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Device failure (General disorders) | 1 | 0 | 0
Medical device complication (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Vaccination site pain (General disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 2 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.